CLINICAL TRIAL: NCT05797883
Title: Clinical Study on the Efficacy and Safety of FOLFOX/FOLFIRI± Targeted Drug Regimen Containing Levofolinic Acid (Zuoyu ®) in the Treatment of Unresectable or Metastatic Colorectal Cancer
Brief Title: FOLFOX/FOLFIRI Containing Levofolinic Acid (Zuoyu ®) in the Treatment of Unresectable or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Chief physician, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-ZY-002
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-01

CONDITIONS: Unresectable or Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX/FOLFIRI (Experimental): q2w, after 8 cycles of medication or patient intolerance or disease progression;
  Interventions: Drug: FOLFOX/FOLFIRI

INTERVENTIONS:
Drug: FOLFOX/FOLFIRI — mFOLFOX6 ：oxaliplatin 85mg/m² IV infusion 2h d1, 5-FU 400mg/m² push d1, Then 5-FU 1200mg/(m2▪d)×2d+Levofolinic Acid 200mg/m² continuous mixed infusion for 46-48h (total 5-FU 2400mg/m²); FOLFIRI ：Irinotecan 180mg/m ² static pulse infusion 30min~90min d1, 5-FU 400mg/m² push d1, Then 5-FU 1200mg/(m2▪d)×2d+ Levofolinic Acid 200mg/m² continuous mixed infusion for 46-48h (total 5-FU 2400mg/m²); The combination of cetuximab/bevacizumab and other targeted agents depends on the patient.

SUMMARY:
To observe and evaluate the efficacy and safety of FOLFOX/FOLFIRI± target-directed regimen containing Levofolinic Acid (Zuoyu ®) in first-line treatment of unresectable or metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years old;
* Patients with histopathologically confirmed unresectable or metastatic colorectal cancer who have not previously received chemotherapy or targeted therapy for unresectable or metastatic lesions;
* Have at least one measurable lesion according to RECIST 1.1 standards;
* ECOG PS score: 0-2;
* Expected survival greater than 3 months;
* Routine blood routine, liver and kidney function, electrocardiogram and other routine tests were basically normal, no contraindications of chemotherapy;
* The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up visits;
* Researchers believe treatment can benefit.

Exclusion Criteria:

* A proven allergy to the test drug and/or its excipients;
* Pregnant or lactating women;
* Patients judged by the investigator to be unsuitable for inclusion in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The proportion of patients whose best overall response (BOR) is complete response (CR) or partial response (PR) assessed by iRECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2years
  The date from random to the first occurrence of disease progression or death from any cause, whichever comes first
Disease control rate (DCR) | 2years
  The proportion of patients whose BOR is CR, PR, and stable disease (SD) assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital & Institute, Shenyang, Liaoning, China